CLINICAL TRIAL: NCT01288690
Title: Stress Reduction in Middle Eastern Refugees
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSU082810B3F
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Refugees; Trauma; Narrative; Exposure; Middle East; Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Narration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait List Control (No Intervention): This condition is a wait-list control and receives no intervention during the study period, but is offered treatment after the final assessment.
- Narrative Exposure Therapy (Experimental): Patients in this condition receive 3 sessions of Narrative Exposure Therapy
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — 3, 1-1/2 hour sessions, individual, meeting weekly.
  Arms: Narrative Exposure Therapy

SUMMARY:
This interventional, randomized controlled study tests the effects of a a brief psychological intervention (Narrative Exposure Therapy) against a wait list control group among refugees who have experienced trauma and have some symptoms of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Refugees from the Middle East, and possible from Africa, who have experienced conflict-related trauma, have symptoms of PTSD, and speak either Arabic or English

Exclusion Criteria:

* Currently received exposure therapy for PTSD
* Planning to leave area in next 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress disorder symptoms: Harvard Trauma Questionnaire | Baseline to 4 months.
  The number and severity of post traumatic stress disorder symptoms will be assessed using an Arabic adaptation of the Harvard Trauma Questionnaire.
  The Harvard Trauma Questionnaire will be administered at baseline prior to randomization and 4 months from baseline (about three months from last intervention session). Questions assess symptoms over the preceding one week.

SECONDARY OUTCOMES:
Physical symptoms: Patient Health Questionnaire | Baseline to 4 months
  Physical symptoms will be assessed using an Arabic translation of the Patient Health Questionnaire at baseline prior to randomization, and 4 months from baseline (about three months from last intervention session). Questions assess symptoms over the preceding 4 weeks.
Depression symptoms: Beck Depression Inventory II | Baseline to 4 months.
  Depression symptoms will be assessed using an Arabic translation of the Beck Depression Inventory II. The scale will be administered at baseline prior to randomization, and 4 months from baseline (about three months from last intervention session). The questions assess symptoms over the preceding two weeks.
Quality of sleep: Karolinska Institute Sleep Questionnaire | Baseline to 4 months
  Quality of sleep will be assessed using an Arabic translation of five items from the Karolinska Institute Sleep Questionnaire. The scale will be administered at baseline prior to randomization, and 4 months from baseline (about three months from last intervention session). The questions don't specify a time frame for the symptoms.
Daily functioning | Baseline to 4 months
  Daily functioning is assessed using 8 items developed by the Primary Investigator in collaboration with other colleagues. The items assess areas such as spending time with family and friends, utilizing health, immigration, language, and employment services, and participating in religious and social activities. The scale will be administered at baseline prior to randomization, and 4 months from baseline (about three months from last intervention session).The questions assess functioning over the preceding 4 weeks.
Post traumatic growth: Post Traumatic Growth Inventory | Baseline to 4 months
  Positive and growth outcomes sometimes experienced by people who have experienced traumatic events will be assessed using an Arabic translation of the Post Traumatic Growth Inventory. The scale will be administered at baseline prior to randomization, and 4 months from baseline (about three months from last intervention session). The questions do not specify a time frame.
General Psychological Well-being: WHO Well-being Index | Baseline to 4 months
  Markers of mental well-being such as positive mood, vitality and interest will be assessed using the Arabic version of the World Health Organization's Well-being Index. The scale will be administered at baseline prior to randomization, and 4 months from baseline (about three months from last intervention session). The questions assess functioning in the preceding two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Lumley, Ph.D, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States